CLINICAL TRIAL: NCT03621527
Title: Efficacy of Fluoroscopy-guided Epidural Anesthesia for Osteoporotic Vertebral Compression Fracture Treated by Percutaneous Vertebroplasty
Acronym: VTB EPI-AL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6833
Record Dates: First submitted 2018-06-07; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-06

CONDITIONS: Vertebral Compression Fractures in Osteoporotic Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (Active Comparator): For each vertebra treated: 10 ml of lidocaine hydrochloride 1% are applied to the skin and the lower structures including the periosteum.
  An additional, anesthesia combined with intravenous analgesia by remifentanil is provided and adapted to the patients needs during the whole procedure
  Interventions: Other: anesthesia combined with intravenous analgesia by remifentanil
- Epidural group (Experimental): Fluoroscopy-guided epidural anesthesiaI is the identification of the epidural space using fluoroscopy and the injection of a small quantity of contrast medium or air.
  According to patient's height, 10-15 ml of lidocaine hydrochloride 1% are injected by the radiologist into the epidural space.
  An additional, anesthesia combined with intravenous analgesia by remifentanil is provided and adapted to the patients needs during the whole procedure
  Interventions: Other: fluoroscopy-guided epidural anesthesia

INTERVENTIONS:
Other: anesthesia combined with intravenous analgesia by remifentanil — intravenous analgesia by remifentanil is provided and adapted to the patients' needs during the whole procedure
  Arms: Standard group
Other: fluoroscopy-guided epidural anesthesia — Identification of the epidural space using fluoroscopy and the injection of a small quantity of contrast medium or air. An additional, anesthesia combined with intravenous analgesia by remifentanil is provided and adapted to the patients needs during the whole procedure
  Arms: Epidural group

SUMMARY:
Vertebral compression fractures in osteoporotic patients is a major healthcare problem. Percutaneous vertebroplasty is commonly used to restore stability of the vertebra and to alleviate pain. However, the anesthetic techniques commonly used during these procedures such general anesthesia or a combination of local anesthesia and sedation are not satisfying as they are associated either with side effects or insufficient pain reduction.

This study compares the standard procedure of local anesthesia to a new technique of fluoroscopy-guided epidural anesthesia carried out by the radiologist.

The investigator's hypothesis is that fluoroscopy-guided epidural anesthesia

* provides better pain relief during the injection of high viscosity cement
* and thus, reduces the need of additional intravenous analgesia by remifentanil (morphine analogue)
* minimizes remifentanil potential adverse effects such as respiratory depression, hypoxemia, pruritus and nausea
* improves working conditions and satisfaction of the radiologist
* improves the global satisfaction of the patient

It is a monocentric, prospective, comparative and randomized study.

ELIGIBILITY:
Inclusion Criteria:

* - Two osteoporotic vertebra compression fractures in the low thoracic or lumbar spine
* men and women > 18 years old
* patients with healthcare insurance
* signed and dated informed consent

Exclusion Criteria:

* men and women < 18 years
* pregnant or breastfeeding women
* patients under trusteeship or guardianship or patients under the protection of court
* bad comprehension or cooperation
* bleeding disorders
* local or general infection
* intracerebral or severe cardiac affections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-03 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Morphine used in the procedure | 1 day
  Maximal target dose of remifentanil used during the procedure to obtain a satisfactory pain reduction during cement injection

CONTACTS AND LOCATIONS:
Overall Officials: Thi Mai BERNEMANN, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No